CLINICAL TRIAL: NCT02507635
Title: In Vivo Anti-inflammatory Effect of H1 Antihistamines in Allergic Rhinitis
Brief Title: Anti-inflammatory H1 Antihistamines Allergic Rhinitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Stefan Cristian Vesa, Assistant professor, Iuliu Hatieganu University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 535
Record Dates: First submitted 2015-07-17; First posted 2015-07-24 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Allergic Rhinitis
Keywords: cytokines; persistent allergic rhinitis; H1 antihistamines
MeSH Terms: conditions — Rhinitis, Allergic | interventions — levocetirizine; desloratadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- healthy volunteers (No Intervention): healthy volunteers
- Desloratadine (Active Comparator): patients with allergic rhinitis under treatment with Desloratadine 5 mg/day, 4 weeks
  Interventions: Drug: Desloratadine
- Levocetirizine (Active Comparator): patients with allergic rhinitis under treatment with Levocetirizine 5 mg/day, 4 weeks
  Interventions: Drug: Levocetirizine

INTERVENTIONS:
Drug: Levocetirizine — administration of Levocetirizine 5 mg/day for 4 weeks
  Other Names: Xyzal
  Arms: Levocetirizine
Drug: Desloratadine — administration of Desloratadine 5 mg/day for 4 weeks
  Other Names: Aerius
  Arms: Desloratadine

SUMMARY:
The main purpose of the treatment of persistent allergic rhinitis is to improve symptoms and patients' quality of life and prevent the development of asthma. Therapeutic strategies also target a reduction of pro-inflammatory mediators released from activated cells, including mast cells and epithelial cells. The presence of allergic inflammation in nasal mucosa may increase the risk of asthma occurrence, especially in patients with persistent allergic rhinitis. H1 antihistamines are widely recommended in all types of allergic rhinitis, regardless of symptom severity or persistence. They control all of the symptoms, but to a lesser extent nasal congestion. New generation agents, such as levocetirizine and desloratadine, possess anti-inflammatory properties, reducing allergic inflammation.

DETAILED DESCRIPTION:
Allergic rhinitis is characterized by a chronic inflammation of nasal mucosa and represents a risk factor for asthma occurrence. H1 antihistamines reduce the rhinitis' symptoms, but some compounds may have anti-inflammatory properties.

We evaluated the plasmatic level of some cytokines in patients with persistent allergic rhinitis (PAR) and their evolution after 4-week treatment with H1 antihistamines and the risk of asthma after 1.5 year.

Eighty-five patients with PAR and 30 healthy volunteers were included in the study. The patients with PAR were randomly divided into 2 groups: 41 patients treated with desloratadine 5 mg/day and 44 patients under levocetirizine 5 mg/day for 4 weeks.

The clinical evaluation include the presence and severity of allergic rhinitis' symptoms: rhinorrhea, nasal congestion, sneezing, nasal and ocular itching and duration of the disease.

Each symptom was evaluated on scale from 0 to 3 (0=absent, 1=mild, 2=moderate, 3=severe) and after that we calculated the total symptoms score (TSS).

A TSS<6 means a mild rhinitis, while a TSS> 6 represented a moderate severe one.

The patients were clinically evaluated after 1.5 year to determine the possible onset of bronchial asthma.

The biological evaluation means determination of total IgE and plasmatic level of IL-1 beta, IL-6, IL-8 and TNF alpha.

Clinical and biological evaluation were performed before and after treatment

ELIGIBILITY:
Inclusion Criteria:

* persistent allergic rhinitis

Exclusion Criteria:

* the presence of asthma or nasal polyps,
* acute and chronic upper respiratory infections,
* administration of intranasal or systemic corticosteroids or H1 antihistamines in the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2009-02; Primary Completion 2011-11 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
efficacy of H1 antihistamines (patients evaluation) | 4 weeks
  patients evaluation before and after 4-weeks treatment

SECONDARY OUTCOMES:
asthma risk (incidence of asthma in patients with persistent allergic rhinitis after 1.5 years from study inclusion) | 1.5 years
  incidence of asthma in patients with persistent allergic rhinitis after 1.5 years from study inclusion

REFERENCES:
- [Derived] Bocsan CI, Bujor AI, Miron N, Vesa SC, Deleanu D, Buzoianu AD. In Vivo Anti-Inflammatory Effect of H1 Antihistamines in Allergic Rhinitis: A Randomized Clinical Trial. Balkan Med J. 2015 Oct;32(4):352-8. doi: 10.5152/balkanmedj.2015.15884. Epub 2015 Oct 1. PMID 26740893